CLINICAL TRIAL: NCT04722328
Title: Establishment of Prevention and Control System of Central Nervous System Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: 04 CNS infection
Record Dates: First submitted 2021-01-19; First posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2020-11

CONDITIONS: Central Nervous System (CNS) Infection; Encephalitis; Meningitis
Keywords: Central nervous system (CNS) infection; diagnosis; pathogen; Metagenomic next generation sequencing
MeSH Terms: conditions — Infections; Encephalitis; Meningitis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CNS infection
  Interventions: Diagnostic Test: CSF metagenomic next generation sequencing (mNGS)
- Non-CNS infection
  Interventions: Diagnostic Test: CSF metagenomic next generation sequencing (mNGS)

INTERVENTIONS:
Diagnostic Test: CSF metagenomic next generation sequencing (mNGS) — TestCSF routine, biochemical, smear staining (Gram staining, acid fast staining, ink staining), culture and mNGS。
  Other Names: CSF detection: routine, biochemical, smear staining (Gram staining, acid fast staining, ink staining), culture.

SUMMARY:
Central nervous system (CNS) infection is a common nervous system acute and severe disease, mainly manifested as encephalitis, meningitis and meningoencephalitis, but also manifested as brain abscess and brain granuloma et al. The basis for the diagnosis of CNS infection lies in the detection of pathogens from brain parenchyma or cerebellar spinal fluid (CSF). However, CSF is relatively difficult to obtain and the sample size is small, which limits the rapid and definite diagnosis of CNS infection pathogens. In addition, CNS infection usually has non-specific clinical manifestations, so it is difficult to identify the pathogen for about half of CNS infection. Metagenomic next generation sequencing (mNGS) and biochip technology provide new means to identify the pathogens of CNS infection. This study analyzes the incidence and epidemic characteristics of CNS infection in China, to standardize the CSF sample processing process, shorten the detection time, increase the sensitivity and specificity of pathogen detection, reduce the detection cost, identify the common pathogens of CNS infection, and establish a standardized rapid diagnosis system, effective prevention and control system.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspected encephalitis or meningitis; onset time within 1 month; modified Rankin Scale (MRS) < 2 points before onset; informed consent of patients; patients who can not express their personal wishes due to aphasia, disturbance of consciousness and other reasons need to obtain the informed consent of their authorized relatives.

Exclusion Criteria:

* Non.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Criteria for clinical suspected encephalitis: acute or subacute onset, fever before and after the onset, symptoms and signs of brain parenchyma damage, including generalized or focal epilepsy (not related to previous epilepsy), mental and behavioral abnormalities, newly emerging local neurological deficit, disturbance of consciousness, etc.
  Clinical suspected meningitis criteria: acute or subacute onset, with fever, headache, vomiting, disturbance of consciousness and meningeal irritation as the main clinical manifestations, accompanied by cranial nerve and brain parenchyma damage.
Sampling Method: Non-Probability Sample
Enrollment: 715 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of pathogen detection | 1 month

SECONDARY OUTCOMES:
I Identify the common pathogens of CNS infection | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Yingfeng Wu, Study Chair — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
The number, age, gender, diagnosis and outcome of the cases.